CLINICAL TRIAL: NCT00844116
Title: Efficacy of "On Line" Telematic Spirometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PI040727
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; spirometry; Telematic spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Spirometry (Active Comparator): personal spirometry
  Interventions: Device: spirometry
- Telematic Spirometry (Experimental): performed remotely "on line"
  Interventions: Device: spirometry

INTERVENTIONS:
Device: spirometry — Conventional and telematic spirometry

SUMMARY:
The investigators aim to demonstrate that spirometry performed "on line" with a technician in a remote place from the patient has the same efficacy as the one performed personally. As a previous study the investigators analyzed the inter-observer agreement between two pulmonary function technicians from both centers taking part in the study: San Pedro de Alcántara Hospital (Cáceres) and Carlos III hospital (Madrid). The main study will be broad (226 patients derivates from primary care to pneumology consultation), prospective, aleatorized, crossed, blind and controlled. The patients will be aleatorized in two groups: 1) personal spirometry: performed in a conventional way; 2) telematic spirometry: performed remotely "on line". The same pulmonary function technician, who will carry out the spirometries personally, will be located in a nearly room. The technician will control the computer office and the spirometer software in the patients's room with another computer. By means of teleconference, the technician will indicate the patient to start the maneuver. After 20 minutes from the end of the first spirometry, the patients will complete the protocol of the following group. The mean values of FVC, FEV1 and FEV1/FVC, the mean time of spirometry performance, the mean number of spirometric maneuvers performed, are compared between both groups by t proof for paired data. The comparison of the percentage of proofs with non acceptability or reproducibility criteria will be made by X2 test. The analysis will be made blindly. The inter-observer and intra-observer agreement will be evaluated by analysis of intraclass correlation for FVC and FEV1 values.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 70 years.
* Patients referred for pulmonary consultation from primary care center.

Exclusion Criteria:

* Psychophysical incapacity to performed spirometry.
* Informed consent not obtained.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The spirometry performed "on line" with a technician in a remote place from the patient has the same efficacy as the one performed personally and FEV1 and FVC | at the end of the study

SECONDARY OUTCOMES:
Nº total test feasible Nº total of test Percentage of cases excluded(dropouts) for failure to obstain three acceptable and two reproducibles test | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Masa, M.D, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Hospital San Pedro de Alcántara. Servicio Extremeño de Salud, Cáceres, Cáceres, Spain